CLINICAL TRIAL: NCT05275257
Title: Can the Use of Uricap Female, a New Urine Collecting Device, Lead to Better Care for Women > 75+Years With Urinary Incontinence?
Brief Title: Can the Use of Uricap Female Device Lead to Better Care for Women > 75+Years?
Acronym: U-PROTECT
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The study never started due to lack of mutual agreements.
Sponsor: Region Örebro County (Other)
Collaborators: Örebro kommun (Unknown); Kumla kommun (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 274847
Record Dates: First submitted 2022-01-31; First posted 2022-03-11 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Urinary Incontinence; Urinary Tract Infections; Incontinence-associated Dermatitis; Cognition Disorders in Old Age; Behavioral and Psychiatric Symptoms of Dementia
Keywords: Long-Term Nursing Homes; BPSD; Urinary incontinence; Urinary Tract Infections; Cognitive decline/dementia
MeSH Terms: conditions — Urinary Incontinence; Urinary Tract Infections; Behavior; Cognitive Dysfunction; Dementia

STUDY DESIGN:
Intervention Model Description: The uridome is changed daily in the intervention group, while the control group will continue to receive the usual incontinence treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Uricap group (Experimental): the new incontinence device
  Interventions: Device: Use of Uricap Female, a New Urine Collecting Device
- Control group (No Intervention): the usual incontinence care

INTERVENTIONS:
Device: Use of Uricap Female, a New Urine Collecting Device — The uridome is changed daily by trained staff
  Arms: Uricap group

SUMMARY:
The purpose of the study is to evaluate if Uricap Female, an uridome for women, can be used instead of traditional incontinence aids to treat urinary incontinence (UI) among women 75 years and older.

DETAILED DESCRIPTION:
The aim is to improve the care for female patients in long-term nursing homes who suffer from UI and to prevent recurrent urinary tract infections (UTIs).

The project organization consist of researchers within primary care, geriatrics and nursing sciences. The investigators will recruit study participants with UI from long-term nursing homes in Örebro County that will be randomized in an open randomised controlled trial to an intervention or a control group. The intervention will last for 3 months. The study participants will receive a structured medical assessment before and after the intervention, including assessment of the patient's cognitive functions, genital skin status, neuropsychiatric symptoms and quality of life (QoL).

The uridome is changed daily while the control group will receive usual incontinence treatment. The investigators will study the number of UTIs during the intervention period, analyze inflammatory cytokines in urine using OLINK proteomics and ELISA to study inflammation. Health economic analysis will be performed.

The investigators believe that treatment with Uricap Female will be more effective in preventing recurrent UTIs, improve genital skin status, cognitive status and neuropsychiatric symptoms and QoL for the women. This will directly lead to individualised care and less strain on primary care resources.

ELIGIBILITY:
Inclusion Criteria:

* UI that requires incontinence aids
* Suitable anatomy (outer labia cover and protect the Uricap Female cup).

Exclusion Criteria:

* active UTI
* urinary retention (cannot empty the bladder on her own)
* macroscopic hematuria
* prolapse or similar gynecological disorders
* allergy to silicone or latex (the material of Uricap Female)
* short expected survival time

Min Age: 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-04 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
UTIs | 12 weeks
  Frequency of incontinence-associated urinary tract infections (UTIs)

SECONDARY OUTCOMES:
Inflammation | Baseline, week 6, week 12
  Grade of inflammation in the urinary tract tissues (inflammation levels assessed by measuring cytokines in urine)
Genital skin status | Baseline, week12
  Asessed using GLOBIAD (plus M) classification tool, grade of incontinence-associated dermatitis (IAD).
Cognitive status | Baseline, week 12
  The patients' cognitive status and neuropsychiatric symptoms for patients with dementia using Mini Mental State Examination Svensk Revidering (MMSE-SR) scale.
  MMSE-SR is assessed on a scale with the minimum and maximum values: 0-30, where a score >25 are seen as normal cognitive status. Lower scores mean a worse outcome.
QoL | Baseline, week 12
  The quality of life using analog EQ-5D-5L with VAS scale.
  EQ VAS registers the patient's self-rated health in a analog scale with the minimum and maximum values: 0-100 where the endpoints are marked: 100 -"The best health you can imagine" and 0 - "The worst health you can imagine". Lower scores mean a worse outcome.
  The quality of life using EQ-5D-5L.
  EQ-5D assesses the current state of health in five dimensions related to well-being and function; mobility, personal care, regular activities, pain/discomfort and anxiety/depression. Each dimension has five levels from "No problems" to "extreme problems". This results in a single-digit number (from 1 to 5) that expresses the level selected for that dimension. Higher digits/scores mean en worse uotcome.
Health economics | baseline, week 11-12
  Nursing time required for incontinence care (minutes per day)
Behavioural and psychological symptoms | Baseline, week 12
  Neuropsychiatric Inventory (NPI) scale.
  NPI is a scale developed to measure behavioral symptoms in various dementia diseases. NPI is assessed on a scale with the minimum and maximum values: 12-144. Higher scores mean a worse outcome/more severe symptoms.
Neuropsychiatric symptoms in dementia | Baseline, week 12
  Cohen Mansfield Agitation Inventory (CMAI) scale
  CMAI is a scale developed to assess behaviors of older adults living in long-term nursing homes. CMAI is assessed on a scale with the minimum and maximum values: 29-203. Higher scores mean a worse outcome.

OTHER OUTCOMES:
Staff interviews | Baseline, week 12
  Is Uricap Female easy to use and how do the nursing staff assess the new treatment method compared to the usual treatment?

CONTACTS AND LOCATIONS:
Overall Officials: Yvonne Freund-Levi, MD, PhD, Principal Investigator — Region Örebro County/Örebro University
Locations (1):
- Department of Geriatrics, University Hospital Örebro, Örebro, Sweden

IPD SHARING:
Plan to Share IPD: No